CLINICAL TRIAL: NCT06140368
Title: The Effect of Virtual Reality on Pain, Anxiety and Patient Comfort During Trigger Point Injection
Brief Title: Virtual Realityon Pain, Anxiety and Comfort During Trigger Point Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Elif Günay İsmailoğlu, Associate Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BU-SBF-EI-003
Record Dates: First submitted 2023-11-10; First posted 2023-11-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Virtual Reality
Keywords: virtual reality; pain; trigger point injection.; anxiety; comfort
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): During the trigger point injection, patients will be shown videos that the patient wants to watch, such as nature and seaside walks, underwater videos, with music background, through virtual reality glasses for 10 minutes.
  Interventions: Behavioral: virtual reality
- Control group (No Intervention): Patients will not use virtual reality glasses during trigger point injection.

INTERVENTIONS:
Behavioral: virtual reality — During the trigger point injection, patients will be shown videos that the patient wants to watch, such as nature and seaside walks, underwater videos, with music background, through virtual reality glasses for 10 minutes.
  Arms: Experimental group

SUMMARY:
To determine the effects of virtual reality application during trigger point injection on patients' pain, anxiety and comfort levels.This research was planned as a randomized controlled experimental type. The population of the research was planned to include patients who applied to the Algology polyclinic for trigger point injection. The sample of the research will consist of 150 patients who meet the sampling criteria and agree to participate in the research.Inclusion criteria: Trigger point injection applied for the first time, 18 years and over, understand and speak Turkish, understand verbal and written information given.Patients will be divided into two groups: experimental (virtual reality) and control groups.Data will be collected with the Case Report Form, State Anxiety Scale, General Comfort Scale and Visual Analog Scale.Patients' anxiety, comfort and pain levels will be evaluated before and after trigger point injection.

DETAILED DESCRIPTION:
Patients in the experimental group will be shown videos that the patient wants to watch, such as nature and seaside walks, underwater videos, with music background, through virtual reality glasses for 10 minutes.Patients in the control group will continue routine practice.Patients' anxiety, comfort and pain levels will be evaluated before and after trigger point injection.

ELIGIBILITY:
Inclusion Criteria:

* The procedure will be applied for the first time

  * 18 years and over
  * Able to understand and speak Turkish
  * Able to understand verbal and written information given
  * Having good cognitive abilities
  * Without visual or hearing loss
  * Patients who agreed to participate in the study

Exclusion Criteria:

* Those who do not understand or speak Turkish
* Does not understand verbal and written information
* Those with impaired cognitive abilities
* Epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
State Anxiety Scale | 10 minutes after procedure
  The scale developed by Spielberger et al. aims to measure state and trait anxiety levels separately.The scores obtained from the scale vary between 20-80, and the total score between 20-39 indicates mild anxiety, between 40-59 indicates moderate anxiety, and between 60-79 indicates severe anxiety.
General Comfort Scale | 10 minutes after procedure
  The scale, which was developed by Kolcaba in 2006 and has a total of 28 questions as 'Refreshing (9 items), Relaxation (9 items) and Overcoming Problems (10 items), consists of three sub-dimensions.The lowest value that can be taken is 1, which indicates low comfort, and the highest value, 6, indicates high comfort.
Visual Analog Scale | In the middle (10 minutes) of the procedure
  It is aimed to determine the level of pain.0 means no pain and 10 means maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Elif Günay İsmailoğlu, Principal Investigator — Izmir Bakircay University
Locations (1):
- Elif Günay İsmailoğlu, Izmir, Menemen, Turkey (Türkiye)